CLINICAL TRIAL: NCT05476198
Title: A Randomized, Controlled Trial Comparing Preoperative Anxiety Effects of Brachial Plexus Block and General Anesthesia for Orthopedic Upper Extremity Surgery
Brief Title: Brachial Plexus Block vs. General Anesthesia for Anesthesia Anxiety Before Orthopedic Upper Extremity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Sertcakacilar, MD, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2020-36
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Orthopedic Disorder; Anxiety; Upper Extremity Injury; Surgery
Keywords: Brachial plexus block; General anesthesia; Orthopedic surgery; Preoperative anxiety; Upper exremity surgery
MeSH Terms: conditions — Musculoskeletal Diseases; Anxiety Disorders; Arm Injuries | interventions — Brachial Plexus Block; Anesthesia, General

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group BPB (Active Comparator): The investigators performed a brachial plexus block on that patient group for preoperative anxiety
  Interventions: Procedure: Brachial plexus block
- Group GA (Active Comparator): The investigators performed general anesthesia on that patient group for preoperative anxiety
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Brachial plexus block — The effect of brachial plexus block method on preoperative anxiety levels in patients who will undergo orthopedic upper extremity surgery.
  Arms: Group BPB
Procedure: General anesthesia — The effect of general anesthesia method on preoperative anxiety levels in patients who will undergo orthopedic upper extremity surgery.
  Arms: Group GA

SUMMARY:
Surgical procedures and anesthesia applications are situations in which people do not feel safe due to the current vital risks. Anxiety is a natural reaction that occurs in such situations, it manifests itself with worry and fear. Increased anxiety before surgery is associated with pathophysiological responses such as hypertension and dysrhythmia. Intense preoperative anxiety can increase morbidity, the need for anesthetic medication, and postoperative analgesia.

For this reason, many questionnaire studies have been conducted to measure the degree of preoperative anxiety and to reveal its causes. The Amsterdam Preoperative Anxiety and Information Scale (APAIS) test has two parts that measure anxiety and the need for information about anesthesia and surgery. The APAIS-A (anxiety) part is the test that measures strain and shows whether the patient has anxiety about anesthesia or surgery. The APAIS-I (information) part estimates whether the person needs information.

In the literature, the effects of general and spinal anesthesia techniques on preoperative anxiety levels have been compared for some specific surgical methods such as c-sections and perianal region surgeries. However, no study has been reported between peripheral nerve block and general anesthesia techniques.

This study aimed to determine the effects of regional and general anesthesia methods on preoperative anxiety levels and the factors affecting these scores in patients who will undergo upper extremity surgery.

DETAILED DESCRIPTION:
146 patients (ASA I-II-III) aged 18-75 years who were to undergo orthopedic upper extremity surgery were randomized and divided into two groups. 26 patients were dropout for different reasons (60 patients in each of the BPB block and general anesthesia groups). One of the brachial plexus blocks was performed according to the level to be operated on to the BPB group, and general anesthesia was performed on the GA group.

Preoperative anxiety of the patients was measured using the APAIS test. The patients' preoperative anxiety score was the primary outcome measure. Postoperative numerical rating scale values were a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-75
* ASA I-III
* Patients who will undergo orthopedic upper extremity surgery

Exclusion Criteria:

* Clinically known local anesthetic allergy
* Morbid obesity (body mass index> 35 kg m2)
* Clinically diagnosis of opioid, alcohol and substance dependence
* Clinically diagnosis of psychiatric disease
* Coagulopathy
* Patients with ASA IV-V
* Illiterate patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety levels in patients who will undergo orthopedic upper extremity surgery with regional or general anesthesia | Preoperative period at day of surgery
  This will be assessed by the Amsterdam Preoperative Anxiety and Knowledge Scale (APAIS) in the preoperative period.
  The APAIS assessment consists of 6 statements. The measure of agreement with these statements should be graded on a 5-point Likert scale from 1 "not at all" to 5 "extremely." The minimum score is 6, the maximum score is 30. A score of ≥11 identifies anxious patients in clinical practice.

SECONDARY OUTCOMES:
Numerical rating scale (NRS) scores of patients | 24 hours postoperatively
  Numerical rating scale (NRS) at 1, 8, 16, 24th hours. NRS assessment score ranges from 0-10. 0 = no pain 10 = worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data available from the publication date can start. Anxiety and NRS scores will be shared. If requested, data will be shared with anesthesiologists dealing with preoperative anxiety.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Chen YK, Soens MA, Kovacheva VP. Less stress, better success: a scoping review on the effects of anxiety on anesthetic and analgesic consumption. J Anesth. 2022 Aug;36(4):532-553. doi: 10.1007/s00540-022-03081-4. Epub 2022 Jul 2. PMID 35779126
- [Background] Ozturk Inal Z, Gorkem U, Inal HA. Effects of preoperative anxiety on postcesarean delivery pain and analgesic consumption: general versus spinal anesthesia. J Matern Fetal Neonatal Med. 2020 Jan;33(2):191-197. doi: 10.1080/14767058.2018.1487948. Epub 2018 Jul 18. PMID 29886798
- [Background] Maheshwari D, Ismail S. Preoperative anxiety in patients selecting either general or regional anesthesia for elective cesarean section. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):196-200. doi: 10.4103/0970-9185.155148. PMID 25948900
- [Background] Celik F, Edipoglu IS. Evaluation of preoperative anxiety and fear of anesthesia using APAIS score. Eur J Med Res. 2018 Sep 11;23(1):41. doi: 10.1186/s40001-018-0339-4. PMID 30205837